CLINICAL TRIAL: NCT04384380
Title: A Multi-center, Randomized, Open-label, Controlled Trial to Evaluate the Efficacy and Tolerability of Hydroxychloroquine (HCQ) in Adult Patients With Mild to Moderate Coronavirus Disease (COVID-19) Compared to Standard of Care Treatment
Brief Title: Efficacy and Tolerability of Hydroxychloroquine in Adult Patients With COVID-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taoyuan General Hospital (Other Government)
Collaborators: Center for Drug Evaluation, Taiwan (Unknown); Centers for Disease Control, Taiwan (Other Government); Taiwan Food and Drug Administration (Unknown); National Health Research Institutes, Taiwan (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TYGH109014
Record Dates: First submitted 2020-04-07; First posted 2020-05-12 (Actual); Last update posted 2020-08-04 (Actual); Status verified 2020-03

CONDITIONS: Coronavirus Infection
Keywords: COVID-19
MeSH Terms: conditions — Coronavirus Infections; COVID-19 | interventions — Hydroxychloroquine

STUDY DESIGN:
Intervention Model Description: The study will employ an open-label parallel design, to evaluate the efficacy and safety between hydroxychloroquine sulfate (plaquenil) and controlled standard of care treatment. The administration plan of HCQ is 400 mg bid on Day 1 and 200 mg bid for 6 days on Day 2-7. All of the enrolled subjects will receive standard of care. The comparison group will receive standard of care, i.e., supportive treatment for subjects with mild COVID-19 clinical illness.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HCQ in adult Patients with COVID-19 (Experimental): The administration plan of HCQ is 400 mg bid on Day 1 and 200 mg bid for 6 days on Day 2-7.
  Interventions: Drug: Hydroxychloroquine Sulfate 200 MG [Plaquenil]
- standard of care treatment (SOC) (No Intervention): The comparison group will receive standard of care, i.e., supportive treatment for subjects with mild COVID-19 clinical illness.

INTERVENTIONS:
Drug: Hydroxychloroquine Sulfate 200 MG [Plaquenil] — Hydroxychloroquine Sulfate is 400 mg bid on Day 1 and 200 mg bid for 6 days on Day 2-7.
  Other Names: Plaquenil
  Arms: HCQ in adult Patients with COVID-19

SUMMARY:
The effective medical treatment against COVID-19 infection is still unknown. Chloroquine phosphate is a well-known antimalarial drug which has been on the market for many years. Recently, in vitro study shown that Chloroquine is effective at both entry and at post-entry stages of the COVID-19 infection of Vero E6 cells with promising results. Chloroquine is also an immune-modifier and could distribute to the whole body including lung. Also, chloroquine is cheap and safe, and could be a promising agent against COVID-19 infection. However, only hydroxychloroquine (HCQ) with the extra hydroxyl group is available in Taiwan. Therefore, hydroxychloroquine instead become the best choice for the treatment candidate, since it shows higher in vitro potency (EC50) against COVID-19 with lower toxicity while retaining the original effect which compared with chloroquine.

DETAILED DESCRIPTION:
On December 31, 2019, an outbreak of respiratory illness later proved to be caused by a novel coronavirus, officially named Coronavirus Disease 2019 (COVID-19), was notified first in Wuhan, a city of Hubei province, People's Republic of China (PRC). COVID-19 rapidly spreads in China and to other parts of the world. Currently more than 370,000 laboratory-confirmed cases have been reported worldwide, and the case count has been rising daily, and caused a global health emergency. As of March 29, 2020, there were 298 confirmed cases in Taiwan.

This is a multi-center, randomized, open-label, controlled trial to evaluate the efficacy and tolerability of Hydroxychloroquine Sulfate (HCQ) in adult Patients with mild to moderate coronavirus disease (COVID-19) compared to standard of care treatment (SOC). The primary endpoint for the study is to evaluate the efficacy of HCQ, with respect to the time to negatively rRT-PCR assessments from the randomization date up to 14 days. The secondary endpoint is to evaluate the efficacy of HCQ in the aspect of virological assessments and the change of clinical symptoms. In addition, the safety and tolerability of HCQ will be evaluated during treatment period in COVID-19 patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who had fever (central temperature ≥38°C) or acute upper respiratory symptoms and laboratory confirmation (rRT-PCR) for COVID-19, with available same type of upper respiratory tract specimens from screening evaluation to the initial testing within 4 days of initial testing
2. Patients have mild (no pneumonia) to moderate disease (pneumonia without respiratory distress) according to the following World Health Organization (WHO) definition of COVID-19 clinical syndromes:

   * Mild (Mild illness):

   Patients with uncomplicated upper respiratory tract viral infection, may have non-specific symptoms such as fever, fatigue, cough (with or without sputum production), anorexia, malaise, muscle pain, sore throat, dyspnea, nasal congestion, or headache. Rarely, patients may also present with diarrhoea, nausea and vomiting.
   * Moderate (Pneumonia):

   Adult with pneumonia but no signs of severe pneumonia and no need for supplemental oxygen.
3. Willing and able to comply with the study procedure and sign a written informed consent

Exclusion Criteria:

1. Patients with the medical history of hypersensitivity to chloroquine, chloroquinine, or hydroxychloroquine
2. Patients with retinal disease, hearing loss, severe neurological and mental illness
3. Patients with pancreatitis
4. Patients with severe lung, liver (alanine aminotransferase (ALT)/aspartate aminotransferase (AST) elevation more than 3 times the normal upper limit), kidney (estimated glomerular filtration rate [eGFR] <30 mL/min/1.73m2, using the MDRD or CKD-EPI methods), brain, haematological diseases or other important systemic diseases
5. Medical history of uncontrolled but clinically significant abnormal cardiac conduction abnormalities at electrocardiogram (ECG) at screening, any history or evidence of long QT syndrome or QTcF interval >450 msec for males and >470 msec for females (according to Fridericia's correction) at screening
6. Known HIV infection; active hepatitis B or C without concurrent treatment (positive tests for hepatitis B [both HBsAg and HBeAg], or high titer of hepatitis C ribonucleic acid [RNA] >800,000 IU/ml)
7. Uncontrolled and unstable concurrent medical condition including psychiatric disorders and alcohol/substance dependence/abuse that will jeopardize the safety of the patient, interfere with the objectives of the study, or affect the patient compliance with study requirements, as determined by the Investigator
8. Patients with concomitant use of medications that alter the absorption or excretion of hydroxychloroquine
9. Patients were considered to be unable to complete the study, or not suitable for the study judged by Investigators
10. Pregnant or breast-feeding women

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2020-05-31 (Actual); Study Completion 2020-05-31 (Actual)

PRIMARY OUTCOMES:
Time to negatively RT-PCR | 14 days
  To evaluate the efficacy of HCQ, with respect to the time to negatively RT-PCR assessments in COVID-19 patients.

SECONDARY OUTCOMES:
Virologic assessment | 14 days
  To evaluate the efficacy of HCQ in the aspect of virologic assessments in COVID-19 patients
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 28 days
  To evaluate the safety and tolerability of HCQ

CONTACTS AND LOCATIONS:
Overall Officials: Shu-Hsing Cheng, Dr., Principal Investigator — Taoyuan General Hospital, Ministry of Health and Welfare
Locations (1):
- Taoyuan General Hospital, Ministry of Health and Welfare, Taoyuan, Taiwan

IPD SHARING:
Plan to Share IPD: No
The study outcome will be shared with the experts and persons interested in this field.

REFERENCES:
- [Result] Cheng SC, Chang YC, Fan Chiang YL, Chien YC, Cheng M, Yang CH, Huang CH, Hsu YN. First case of Coronavirus Disease 2019 (COVID-19) pneumonia in Taiwan. J Formos Med Assoc. 2020 Mar;119(3):747-751. doi: 10.1016/j.jfma.2020.02.007. Epub 2020 Feb 26. PMID 32113824
- [Result] Huang C, Wang Y, Li X, Ren L, Zhao J, Hu Y, Zhang L, Fan G, Xu J, Gu X, Cheng Z, Yu T, Xia J, Wei Y, Wu W, Xie X, Yin W, Li H, Liu M, Xiao Y, Gao H, Guo L, Xie J, Wang G, Jiang R, Gao Z, Jin Q, Wang J, Cao B. Clinical features of patients infected with 2019 novel coronavirus in Wuhan, China. Lancet. 2020 Feb 15;395(10223):497-506. doi: 10.1016/S0140-6736(20)30183-5. Epub 2020 Jan 24. PMID 31986264
- [Result] Zhang W, Du RH, Li B, Zheng XS, Yang XL, Hu B, Wang YY, Xiao GF, Yan B, Shi ZL, Zhou P. Molecular and serological investigation of 2019-nCoV infected patients: implication of multiple shedding routes. Emerg Microbes Infect. 2020 Feb 17;9(1):386-389. doi: 10.1080/22221751.2020.1729071. eCollection 2020. PMID 32065057
- [Result] Cortegiani A, Ingoglia G, Ippolito M, Giarratano A, Einav S. A systematic review on the efficacy and safety of chloroquine for the treatment of COVID-19. J Crit Care. 2020 Jun;57:279-283. doi: 10.1016/j.jcrc.2020.03.005. Epub 2020 Mar 10. PMID 32173110
- [Result] Gautret P, Lagier JC, Parola P, Hoang VT, Meddeb L, Mailhe M, Doudier B, Courjon J, Giordanengo V, Vieira VE, Tissot Dupont H, Honore S, Colson P, Chabriere E, La Scola B, Rolain JM, Brouqui P, Raoult D. RETRACTED: Hydroxychloroquine and azithromycin as a treatment of COVID-19: results of an open-label non-randomized clinical trial. Int J Antimicrob Agents. 2020 Jul;56(1):105949. doi: 10.1016/j.ijantimicag.2020.105949. Epub 2020 Mar 20. PMID 32205204

DOCUMENTS (1):
  • Study Protocol (2020-03-29): https://cdn.clinicaltrials.gov/large-docs/80/NCT04384380/Prot_000.pdf